CLINICAL TRIAL: NCT06801067
Title: A Single-Arm, Open-Label, Phase 1 Study to Assess Safety and Preliminary Efficacy of Cultivated Multi-Strain Live Bacterial Therapeutic SER-155 for First-Line Treatment of Immunotherapy-Related Enterocolitis
Brief Title: A Study of SER-155 to Treat Diarrhea in People on Immunotherapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-231
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Diarrhea; Enterocolitis
Keywords: Diarrhea; SER-155; Enterocolitis; Memorial Sloan Kettering Cancer Center; 24-231
MeSH Terms: conditions — Diarrhea; Enterocolitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Immune checkpoint inhibitor-related enterocolitis (irEC) (Experimental): Participants with grade 2-3 diarrhea from irEC who have not yet received immunosuppressive therapy for irEC
  Interventions: Biological: SER-155

INTERVENTIONS:
Biological: SER-155 — SER-155 (Cultivated Multi-Strain Live Bacterial Therapeutic, Encapsulated) is an experimental designed ecology of 16 unique, human-commensal bacterial strains encapsulated for oral administration and will be provided by Seres as an investigational drug
  Other Names: Cultivated Multi-Strain Live Bacterial Therapeutic, Encapsulated

SUMMARY:
The purpose of this study is to find out whether SER-155 may be a safe first treatment that causes few or mild side effects for people due to irEC.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Receipt of ICI (single-agent or combination) within the 180 days preceding screening.

Concurrent treatment with cytotoxic chemotherapy or other tumor-directed agents is permitted.

* Grade 2 - 3 diarrhea (i.e., increase of at least 4 bowel movements a day above baseline during the screening window), deemed by the treating provider as likely related to ICI therapy, with or without concomitant symptoms of grade 1 - 2 colitis (e.g.

abdominal pain, bloody or mucoid stools)

* Able to swallow oral medication
* Individuals of childbearing potential willing to use a highly effective method of contraception (failure rate of <1% per year when used consistently and correctly) for 30 days after the last dose of SER-155.
* Willing to provide written informed consent, comply with the protocol, and understand the potential risks and benefits of study enrollment and treatment.

Exclusion Criteria:

* Active GI infection, including untreated viral, bacterial or fungal cause(s) of diarrhea.
* Received immunosuppressive therapies for suspected or confirmed irEC, including systemic corticosteroids (either oral or intravenous) and/or infliximab, vedolizumab or ustekinumab
* Grade 3 colitis symptoms, i.e. severe abdominal pain or peritoneal signs
* Admitted to the hospital for irEC
* Prednisone (or steroid equivalent) dose > 10 mg a day for a non-GI irAE at time of screening
* Pre-existing inflammatory bowel disease (e.g. Crohn's disease or ulcerative colitis) or microscopic colitis
* Pregnant or lactating women
* Any condition that requires ongoing prophylactic or therapeutic antibacterial antibiotics
* Severe neutropenia, as defined by an absolute neutrophil count (ANC) < 500 cells/mm^3, at time of screening
* Treatment with investigational medications used for diarrhea/colitis treatment and microbiome therapeutics within 30 days prior to enrollment
* Known allergy or intolerance to oral vancomycin
* Unable to comply with the protocol requirements
* Any condition that in the opinion of the investigator may increase the risk of study participation and/or may interfere with the interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2027-01-24 (Estimated); Study Completion 2027-01-24 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with treatment-related adverse events of special interest | 1 year
  Proportion of participants with treatment-related adverse events of special interest, i.e. blood stream infection
Proportion of patients with treatment-related adverse events | 1 year
  Proportion of patients with treatment-related adverse events

SECONDARY OUTCOMES:
Proportion of patients with immunosuppressive-free clinical response of irEC (immunotherapy-related enterocolitis) at day 15 | Day 15
  Proportion of patients with immunosuppressive-free clinical response of irEC (immunotherapy-related enterocolitis) at day 15, defined as at least one grade decrease in diarrhea symptoms without the use of immunosuppressive therapy
Proportion of patients with immunosuppressive-free clinical remission of irEC at day 15 | Day 15
  Proportion of patients with immunosuppressive-free clinical remission of irEC at day 15, defined as resolution in diarrhea symptoms (grade 0) without the use of immunosuppressive therapy
Proportion of patients with immunosuppressive-free clinical response of irEC at day 43 | Day 43
  Proportion of patients with immunosuppressive-free clinical response of irEC at day 43
Proportion of patients with immunosuppressive-free clinical remission of irEC at day 43 | Day 43
  Proportion of patients with immunosuppressive-free clinical remission of irEC at day 43
Time to immunosuppressive-free clinical response | 1 year
  Time to immunosuppressive-free clinical response
Time to immunosuppressive-free clinical remission | 1 year
  Time to immunosuppressive-free clinical remission
Number of detectable SER-155 strains at day 15 | Day 15
  Number of detectable SER-155 strains at day 15
Number of detectable SER-155 strains at day 43 | Day 43
  Number of detectable SER-155 strains at day 43

CONTACTS AND LOCATIONS:
Overall Officials: David Faleck, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memoral Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited protocol activity), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org